CLINICAL TRIAL: NCT03303287
Title: School Health Education Program in Pakistan(SHEPP) ; Impact on Lifestyle and Cardio-
Brief Title: School Health Education Program in Pakistan(SHEPP)
Acronym: SHEPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Aysha Almas, Associate professor, Aga Khan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEC_4553
Record Dates: First submitted 2017-09-27; First posted 2017-10-06 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Health Education
Keywords: health education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: : Three schools under the Aga Khan Education Service in Karachi will be included in a two-arm parallel cluster intervention trial. All schools belong to lower to middle income class, at different locations, all having the same school curriculum. Baseline data will be collected from all three schools during a three month period by trained research staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): School health education program in Pakistan(SHEPP): The health education program will be directed towards children, parents and teachers
  Interventions: Behavioral: School health education
- control (No Intervention): usual

INTERVENTIONS:
Behavioral: School health education — School health education program in Pakistan(SHEPP): The health education program will be directed towards children, parents and teachers
  Arms: intervention

SUMMARY:
Pakistan is a developing country and there have been a considerable rise in obesity and hypertension in children in recent years. In this setting a focus on primary prevention of cardiovascular diseases is more cost effective than spending resources on secondary or tertiary prevention,. Primary prevention includes interventions to promote physical activity (> 30 minutes/day in school), healthy dietary habits (decreased consumption of sweetened beverages and snacks, and increased consumption of fruit and vegetables) and health education focusing on cardiovascular risk factors in school children. This would translate into healthier cardiovascular outcomes (eg. less hypertension, dyslipidemia and diabetes) in adult life. The investigators propose a school health education program for Pakistan (SHEPP) for children aged 9-11 years in 3 schools in Karachi for a period of one year. This program will comprise of 140 minutes physical activity/week (including aerobics):30 minutes aerobic PA(30*2=60) + 10 minutes (10*5=50)physical activity in assembly daily+ 1 minute between periods(1*6*5=30) and healthy diet and healthy heart teaching. Additionally teaching will also be given to teachers and parents, who will further reinforce these habits in children. We hypothesise that SHEPP will improve physical activity levels, dietary habits and knowledge about healthy heart in children, will decrease blood pressure, body mass index, waist circumference, at the end of the year. If this healthy behavior is carried on to adult life it will serve as an excellent primary prevention measure. The investigators , later on plan to study long term outcomes after implementation of this intervention.

DETAILED DESCRIPTION:
1.1.Interventions to reduce childhood obesity School based programs have also been introduced as interventions to assess the impact on blood pressure ant weight. In effectiveness trial done by Yin et al on the impact of 8 months after school physical activity programme demonstrated a reduction in percentage body fat, but no effect on blood pressure.(52) Schools have been unable to provide sufficient time and resources for students to meet all the objectives of standard physical education, the concept of "health-related PE".(13)Traditionally, the role of schools in providing and promoting physical activity has been during the school day (eg, PE, recess) and/or on the school campus immediately after school. Trial of Activity for Adolescent Girls (TAAG) is a large-scale randomized trial involving 36 schools at 6 study sites across the United States and sponsored by the National Heart, Lung, and Blood Institute. This large-scale study is examining the effects of a school-community linked intervention on overall physical activity in middle school girls.(53)

Physical activity and behavior of change theory The effectiveness of physical activity interventions would benefit from a better understanding of this behavior. (54) Theory of planned behavior has demonstrated usefulness in studies of health-related behavior.(55) Only children's intention and self-identity as a result of their cognition is related to participation in physical activity to some extent(56). This suggests that educational strategies aimed at increasing children's motivation remainan important strategy to promote physical activity. Physical activity interventions have been done focusing on designing interventions to overcome cultural, socioeconomic barriers in performing physical activity based on psychosocial cognitive theory.(57)

A number of carefully designed studies incorporating health-related PE concepts and physical activity in PE classes have been conducted. Dietary or physical activity behavior produce a significant and clinically meaningful reduction in body mass index status of children and adolescents in preventing obesity (58, 59) Alternatively behavioral prevention and situational prevention elements have been combined to increase physical activity, decrease the consumption of sugar-sweetened beverages, and decrease time spent with screen media(60).

Studies reporting positive outcomes implemented physical activity sessions that lasted at least 30 min d(-1)?. Several studies showed that children are most active in the first 10-15 min. The existence or installation of playground markings or fixed play equipment had no effect, whereas the presence or addition of portable play equipment was positively correlated with moderate-to-vigorous physical activity.

Role of Parents and Teachers One of the interventions in promoting healthy lifestyle in children is focusing on children, parents and teachers simultaneously by introducing learning sessions and materials for healthy lifestyle.(32, 61)Teacher training may be a key element for successful interventions. To overcome time constraints, a suggested solution is to integrate physical activity into daily routines and other areas of the preschool curriculum.(62)Additionally parental barriers are associated with the time that children spend in both active and sedentary pursuits.(63) Knowledge about risk factors for obesity and myocardial infarction is suboptimal in Pakistani adults(64).Only 42% adult students had a good level of knowledge of modifiable risk factors of heart disease among patients with acute myocardial infarction in Karachi.(65)Health education on physical activity and healthy diet using multiple level intervention is essential to be given at schools.

1.2 Rationale Dietary behaviors, physical activity and sedentary lifestyle are independent predictors of overweight and higher BMI among Pakistani primary school children.(66) Your study does not focus on preschool children so it is better to write about school children. Children skipping breakfast (8%), eating fast food and snacks ≥once a week (43%) and being involved in sedentary lifestyle>one hour a day (49%) were significantly more likely to be overweight and obese while those participating in physical activity>twice a week (53%) were significantly less likely to be overweight and obese.(67) Approximately 85% of the students had a predominantly sedentary life style, due to tuitions, television viewing or internet surfing or indoor games like play stations in affluent schools of Karachi.(68)Most public sector schools do not have designated physical trainers to encourage physical activity in school children. Additionally unhealthy food including fast food, sugar sweetened beverages are commonly available in the school canteens. Furthermore the television watching and computers have added to physical inactivity making the children more sedentary. Most schools do not have any health education curriculum which could be taught to children and no such trial has been conducted in Pakistan A feasibility study using a similar design was done including 276 children, in which 60 % spent > 3 hours daily in watching TV or working on computer. It was conducted in four public sector schools in Karachi. However due to limited length of intervention of 20 weeks, clear benefits on cardiovascular outcomes like blood pressure could not be observed (unpublished data).Additionally incorporating 30 min physical activity was a challenging task and was not sustainable. Maybe this is something for the summary since you already have said it :Schools are probably the most pragmatic place where such shifts in lifestyle can be incorporated in adolescents.( figure 1) Strategies for promoting physical activity at school level have been tested worldwide , however not at large in Pakistan. Strategies need to be built in on large scale in adolescents, which can be incorporated within their school boundry and time limitations. A multipronged approach involving children, parents and teachers simultaneously is needed in school setup to make it more successful. Using a multilevel approach to childhood obesity prevention including staff, parents, and community partners is beneficial.(69) )

1.3.Main aim The main aim of the study is to incorporate a healthy lifestyle in children in terms of increased physical activity, healthier dietary habits, and basic health education. The hypothesis is that the programme will increase the level of physical activity not only at school time but also at leisure time, increase the healthy dietary habits and have an effect on cardiovascular outcomes.

1.4 Research Questions 1.4a. Research question I

* What is the effect of a 10 months school health education program in Pakistan(SHEPP): vs routine physical activity levels (in school, out of school, moderate to vigorous physical activity and sedentary time) in school children ? 1.4b. Research questions II
* What is the effect of a 10 months school health education program in Pakistan(SHEPP): vs routine on intake of fruits and vegetable, sugar sweetened beverages and snacks taken/day in school children ? 1.4c.Research question III
* What is the effect of a 10 months school health education program in Pakistan(SHEPP)vs routine on cardio metabolic risk factors; systolic blood pressure, diastolic blood pressure, body mass index and waist circumference and body fat percentage in school children?

1.5. Objectives 1.5a. Objective I

* To compare the effect of a 10 months school health education program in Pakistan(SHEPP): vs routine on physical activity levels (in school, out of school, moderate to vigorous physical activity and sedentary time) in school children 1.5b. Objective II
* To compare the effect of a 10 months school health education program in Pakistan(SHEPP): vs routine on intake of fruits and vegetable, sugar sweetened beverage and snacks taken/day in school children 1.5c.Objective III
* To compare the effect of a 10 months school health education program in Pakistan(SHEPP)vs routine on cardio metabolic risk factors; systolic blood pressure, diastolic blood pressure, body mass index and waist circumference and body fat percentage in school children

  2. Methods 2.1 Study Design Study design and participants: Three schools under the Aga Khan Education Service in Karachi will be included in a two-arm parallel cluster intervention trial. All schools belong to lower to middle income class, at different locations, all having the same school curriculum. Baseline data will be collected from all three schools during a three month period by trained research staff. This would comprise of data on sociodemographic factors, FFQ for diet, youth physical activity questionnaire for physical activity, blood pressure ,weight, height and waist circumference, body fat percentage measurements using validated instruments. Each school will then be assigned to intervention or control (intervention in one school , and control in 2 schools). All children aged 8-11 years enrolled in these schools will be included. The rationale for this is that it is the period 8-11 years age where physical activity starts to decline mainly in girls.(70) Follow up will be done after 10 months of intervention. Ten months cutoff has been chosen as benefits on cardiovascular risk factors are more pronounced at 10 month follow-up.(39)

2.2 Study Setting

Schools under the Aga Khan Education Service will be selected since they are all part of Aga Khan Development network. These are:

1. Aga Khan School, Kharadhar
2. Aga Khan School, Garden
3. Sultan Mohamed Shah Aga Khan School, Karachi The reason for selection of these school is that they follow a uniform curriculum across the school system. Additionally since they are apart of the Aga Khan Development network, it would be more practical to work with them. All schools are located in urban Karachi and Hyderabad. They have ample space to conduct physical activity sessions, auditoriums and discussion room. Each school has approximately 2000 students, both boys and girls. Each school comprises of 10 levels of classes with 3-4 sections. The study is expected to be completed in 18 months to 20 months.

Intervention School health education program in Pakistan(SHEPP): The health education program will be directed towards children, parents and teachers. The basis of designing such intervention is to overcome cultural, socioeconomic barriers in performing physical activity and is based on psychosocial cognitive theory.(57)The primary focus will be the children.(figure II) Children 4. Programmed physical activity 140 minutes / week will be targeted. i. 30 minutes twice a week will be delivered by teachers trained by expert physical trainers. It would comprise of warm up, moderate to vigorous physical activity and cool down(71).(30*2=60 min/week). These sessions will be lead by the school physical trainer under supervision of an expert physical trainer (trained in aerobics) Different exercises is introduced every month and discussions with students will be done by the research team as well. A manual will be built to keep uniformity in the interventions. This has been previously tested(71) ii. 10 minutes physical activity daily during assembly(10*5=50 minutes/week) iii. 1 minute between class warm up. (1*6*5=30 minutes/week) Children will be encouraged to perform brake time physical activity by selecting leaders within a class group(who will facilitate such PA in brake time)

* Perform such PA in leisure time 4 times a week(atleast half an hour)
* Before class exercises(2 minutes between periods)
* Decrease levels of sedentary behavior(not more than hour) 5. Healthy diet teaching will be given to children by a trained nutritionist. Healthy diet is based on food pyramid.(72)There would be three sessions in all of one hour duration i. Encouragement to increase fruits and vegetables intake serving in a day ii. Encouragement to avoid sugar sweetened beverages iii. Encouragement to avoid fast food items 6. Healthy heart teaching will be given by a trained physician. This would comprise of total 7 sessions (one hour each). The study material for the children will be adapted from "my heart" (www.bookgroup.org.pk, Children health fund). This material has been pilot tested earlier in schools. It has basic information about heart. (AppendixA)
* Heart
* Blockage of arteries
* Riskfactors for blockage
* Diet
* Physical activity
* Smoking and smokeless tobacco
* Hand and dental Hygiene
* Anger mangement Parents Group health education to parents-will be done by the team of trained nutritionist, physician and teachers. Teachers will be trained to teach parents. This will be done on weekends in large class format. It would comprise of one hour each.

  1. Health problems in Pakistan
  2. Physical activity as a preventive measure
  3. Healthy diet as a preventive measure Parents will then reinforce these habits in their children and will ask them atleast twice a week.(Did ypu do physical activity at school and home?Did you have atleast one fruit or vegetable today?) Teachers The teachers will be trained by a team of experts including a physician, a nutritionist and a physical activity expert. A teachers guide will be developed.(Appendix B)This comprises of
* Heart
* Blockage of arteries
* Risk factors for blockage
* Diet
* Physical activity
* Smoking and smokeless tobacco
* Hand and dental Hygiene
* Anger management The teachers will then reinforce about healthy physical activity and diet in class once /week (did you do physical activity at home and school?How many times did you take fruits and vegatables?).

ELIGIBILITY:
Inclusion Criteria:

* All children aged 8-11 years enrolled in the schools.

Exclusion Criteria:

* Any child or adolescent suffering from any physical disability

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
increase in Minutes spent in school, out of school in physical activity | 10 months
  • Physical activity levels(in school, out of school, moderate to vigorous physical activity and sedentary time) assessed by number of minutes spent in physical activity

SECONDARY OUTCOMES:
decrease in blood pressure in mm | 10 months
  blood pressure
decrease in BMI in kg/m2 | 10 months
  BMI= weight in kg/height in meter square
increase in Number of fruits and vegetable/ decrease in sweetened beverages in a day | 10 months
  • Dietary patterns in terms of fruits and vegetable serving, sweetened beverages and snacks/day
Decrease in waist circumference in cm | 10 months
  Decrease in waist circumference in cm

CONTACTS AND LOCATIONS:
Overall Officials: Aysha Almas, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan Schools, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Almas A, Iqbal R, Ghani A, Samad Z, Sabir S, Kazmi K. School Health Education Program in Pakistan (SHEPP): findings from a feasibility trial in pre-adolescent school children from a lower middle-income country. Pilot Feasibility Stud. 2023 Jul 17;9(1):123. doi: 10.1186/s40814-023-01344-9. PMID 37461089
- [Derived] Almas A, Iqbal R, Sabir S, Ghani A, Kazmi K. School health education program in Pakistan (SHEPP)-a threefold health education feasibility trial in schoolchildren from a lower-middle-income country. Pilot Feasibility Stud. 2020 Jun 8;6:80. doi: 10.1186/s40814-020-00625-x. eCollection 2020. PMID 32523724